

NCT Number: NCT04667338

Title: Observational, Multicentre, Cross-sectional Study to Describe Diagnosis and

Treatment Patterns in Narcolepsy Patients in Real Life Practice in Spain

Study Number: TAK-994-5001 (Narcolepsy-5001)

Document Version and Date: 1.0 (19 January 2023)

Certain information within this document has been redacted (ie, specific content is masked e info irreversibly from view) to protect either personally identifiable information or company

confidential information.



PROTOCOL NUMBER: Narcolepsy-5001

OBSERVATIONAL, MULTICENTRE, CROSS-SECTIONAL STUDY TO DESCRIBE DIAGNOSIS AND TREATMENT PATTERNS IN NARCOLEPSY PATIENTS IN REAL LIFE PRACTICE IN SPAIN

AUTHOR:

**VERSION NUMBER AND DATE: 1.0; 19JAN2023** 

Document: SAP SOMNUS

Author: Version Number: 1.0

Version Date: [19JAN2023]

Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



Statistical Analysis Plan Page 2 of 80

# STATISTICAL ANALYSIS PLAN SIGNATURE PAGE

Statistical Analysis Plan V 2.0 for Protocol Narcolepsy-5001.

| | Name | Signature | Date |
|--------------|----------------|--------------|------|
| Author: | | | |
| Position: | | | |
| Company: | IQVIA | | |
| | | 070 | |
| | Name | Signature | Date |
| | Name | Signature | Date |
| Approved By: | | Thing cial | |
| Position: | | OINE, | ' |
| Company: | | COICH | |
| | 70- | | |
| Approved By: | 1.0 | | |
| Position: | | | |
| Company: | Takeda Farmacé | utica España | |

Document: SAP SOMNUS

Version Date: [23SEP2022]

Version Number:

1.0

Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Oct2021



# **MODIFICATION HISTORY**

| Unique | Date of the | Author | Significant Changes from |
|---|---|---|---|
| Identifier | Document | | Previous Authorized Version |
| for this | Version | | |
| Version | | | |
| Draft 1.0 | 24 MAY 2022 | | Not Applicable – First draft |
| Draft 2.0 | 23 SEP 2022 | | Restructuring of the tables and add models |
| Draft 3.0 | 24NOV 2022 | | Reviewing comments from Study |
| | | Sicilo | Coordinators |
| Draft 4.0 | 18JAN2023 | alline | No significant modifications |

Document: SAP SOMNUS

Template No.: RWI\_TP\_BIOS0013 Revision 2

Author: Version Number: 1.0 Version Date: [19JAN2023]

Reference: RWI\_WI\_BIOS0015



# **TABLE OF CONTENTS**

| P | <b>ABBR</b> | REVIATIONS6 |
|---|---|---|
| | | ODUCTION |
| \$ | STUD | Y OBJECTIVES |
| _ | 3.1 | Primary Objectives |
| _ | 3.2 | Secondary Objectives |
| | 3.3 | Exploratory Objectives |
| 5 | STUD | Y DESIGN9 |
| 4 | 4.1 | General Description 9 |
| 4 | 4.2 | Schedule of Events 10 |
| 4 | 4.3 | Changes to Analysis from Protocol |
| 1 | PLAN | NED ANALYSES |
| 4 | 5.1 | Interim Analysis |
| 5 | 5.2 | Final Analysis |
| A | ANAI | YSIS SETS11 |
| 6 | 5.1 | Y DESIGN 9 General Description 9 Schedule of Events 10 Changes to Analysis from Protocol 10 NED ANALYSES 10 Interim Analysis 10 Final Analysis 10 All Subjects Enrolled Set [ENR] 11 6.1.1 Inclusion criteria 11 6.1.2 Exclusion criteria 11 Sefety Analysis Set [SAE] 12 |
| | | 6.1.1 Inclusion criteria |
| | | 6.1.2 Exclusion criteria |
| 6 | 5.2 | Safety Analysis Set [SAF] 12 CRAL CONSIDERATIONS 12 |
| | GENE | CRAL CONSIDERATIONS12 |
| | 7.1 | Windowing Conventions |
| 7 | 7.2 | Collected Variables and Measures |
| | | 7.2.1 Primary endpoint |
| | | 7.2.2 Secondary endpoints |
| | | 7.2.3 Exploratory endpoints |
| | | 7.2.4 Other analysis |
| | 7.3 | Software Version |
| 5 | STAT | ISTICAL CONSIDERATIONS |
| 8 | 3.1 | Statistical Tests and Confidence Intervals |
| 8 | 3.2 | Adjustments for Covariates and Factors to be Included in Analyses |
| 8 | 3.3 | Missing data |
| 8 | 3.4 | Examination of Subgroups |
| 8 | 3.5 | Derived variables |
| | OUTP | PUT PRESENTATIONS |
| 1 | DISPO | OSITION AND WITHDRAWALS20 |

Template No.: RWI\_TP\_BIOS0013 Revision 2

Effective Date: 15Oct2021

Author:


Version Date:

1.0

Reference: RWI\_WI\_BIOS0015

[19JAN2023]



| 11. | <b>DEM</b> ( | OGRAPHIC AND OTHER BASELINE CHARACTERISTICS | 20 |
|---|---|---|---|
| <b>12.</b> | <b>MEDI</b> | CAL HISTORY | 21 |
| <b>13.</b> | CONC | COMITANT ILLNESSES | 21 |
| 14. | <b>MEDI</b> | [CATIONS | 22 |
| <b>15.</b> | <b>PATI</b> | ENT REPORTED OUTCOMES (PRO) | 22 |
| | 15.1 | WPAI-GH | 22 |
| | 15.2 | EQ-5D | 23 |
| | 15.3 | SSCI-8 | 23 |
| | 15.4 | TSQM-9 | 23 |
| <b>16.</b> | SAFE | TY OUTCOMES | 24 |
| <b>17.</b> | | RENCES | |
| <b>18.</b> | <b>APPE</b> | NDIX 1. PROGRAMMING CONVENTIONS FOR OUTPUTS | |
| | 18.1 | Inclusion-exclusion criteria | 27 |
| | 18.2 | Demographic and baseline characteristics | 28 |
| | 18.3 | Diagnosis of narcolepsy | 31 |
| | 18.4 | Demographic and baseline characteristics Diagnosis of narcolepsy Comorbidities Treatment patterns | 35 |
| | 18.5 | Treatment patterns | 42 |
| | 18.6 | Direct and indirect healthcare resources utilization | 49 |
| | | 18.6.1 Healthcare resources in the last 12 months prior to study visit | 49 |
| | | 18.6.2 Healthcare resources before diagnosis of narcolepsy | 58 |
| | 18.7 | Patient Reported Outcomes (PRO) | |
| | | 18.7.1 Health-Related Quality of Life (HRQoL) | 64 |
| | | 18.7.2 Perception of stigma | |
| | | 18.7.3 Treatment satisfaction | 66 |
| | 18.8 | Factors related to healthcare resources utilization, quality of life, stigma | |
| | | and satisfaction. | 67 |
| | 18.9 | Proportion of patients with narcolepsy diagnosed and managed in public | |
| | | hospitals | 71 |
| | 18.10 | Sociodemographic and clinical characteristics of patients with narcolepsy | |
| | | according to treated and untreated patients. | |
| | 18.11 | Adverse drug reaction associated to narcolepsy treatments | 75 |
| <b>19.</b> | ANNE | X | 76 |

Document: SAP SOMNUS

Author:


1.0


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



#### 1. ABBREVIATIONS

AE: Adverse Event

ADR: Adverse Drug Reaction AHI: Apnea-hypopnea index CCI: Charlson Comorbidity Index

CRF: Case Report Form CSF: Cerebrospinal fluid

eCRF: electronic Case Report Form EO-5D: EuroQol five-dimensions .atness Test
.aents
.asy type 1
.arcolepsy type 2
Polysomnography
Patient Recorded Outcomes
Rapid eye movements
'afety Analysis Set
atistical Analysis
stained ^ ENR: ESS: HLA: HRQoL: MSLT: MVAs:

MWT:

NMAs: NT1: NT2: PSG:

PRO:

REM: SAF: SAP:

SART:

SD: Standard Deviation

SSCI: 8-item Stigma Scale for Chronic Illness

SOREMPs: Sleep-onset REM periods

TSQM-9: Treatment Satisfaction Questionnaire Medication

WPAI-GH: Work Productivity and Activity Impairment Questionnaire General

Document: SAP SOMNUS


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI WI BIOS0015



#### 2. INTRODUCTION

Statistical Analysis Plan

This statistical analysis plan (SAP) describes the rules and conventions to be used in the presentation and analysis of management and treatment patterns of narcolepsy in adults' patients in real world practice in Spain. It describes the data to be summarized and analyzed, including specifics of the statistical analyses to be performed.

This statistical analysis plan (SAP) is based on protocol version 2.0, dated 20<sup>th</sup> December 2021 and Offinercial Use of box amendments 1 and case report forms (CRFs) version 3.0, dated 19th January 2022.

#### 3. STUDY OBJECTIVES

#### 3.1 **Primary Objectives**

The primary objective of the study is:

To describe the treatment patterns (pharmacological and non-pharmacological)

- o in patients with narcolepsy between different subgroups, including:
  - Patients with and without cataplexy \* (*Note: Patients with narcolepsy type 1 and type 2*)

Patients treated and naïve-treatment patients (Note: not pharmacological treatments)

- \* New terminology regarding type of narcolepsy has been consensed:
  - Patients with narcolepsy Type 1 are those patients with cataplexy
  - Patients with narcolepsy Type 1 are those patients without cataplexy

This new terminology has been applied in all this document accordingly

Document: SAP SOMNUS

Template No.: RWI\_TP\_BIOS0013 Revision 2

Version Number: 1.0


Reference: RWI WI BIOS0015



#### 3.2 **Secondary Objectives**

The secondary objectives are:

Statistical Analysis Plan

- 1. To characterize sociodemographic and clinical characteristics of patients with narcolepsy and compare it between treated and untreated patients in Spain.
- 2. To describe specialists involved in diagnosis of patients with narcolepsy in Spain.
- 3. To describe diagnosis processes used in real-world as described in patients' medical records in Spain.
- 4. To evaluate and describe effectiveness (treatment outcomes) of the currently used narcolepsy treatments in the study period in Spain.
- 5. To estimate direct costs associated with narcolepsy patients in Spain, in terms of treatment, number of visits, hospitalization, and additional resources within the last 12 months before study visit.
- 6. To estimate indirect costs associated with narcolepsy patients in Spain, using the Work Productivity and Activity Impairment Questionnaire General (WPAI-GH).
- 7. To describe the health-related quality of life (HRQoL) of patients with narcolepsy in Spain using the EQ-5D Questionnaire.
- 8. To assess the perception of stigma of patients with narcolepsy in Spain using the 8-item Stigma Scale for Chronic Illness (SSCI-8).
- 9. To describe treatment satisfaction of patients with narcolepsy in Spain using the Treatment Satisfaction Questionnaire Medication (TSQM-9).
- 10. To describe the burden of illness in terms of associated comorbidities and associated disorders in the last 12 months.
- 11. To describe adverse drug reaction (ADR) associated to narcolepsy treatments

#### 3.3 **Exploratory Objectives**

The exploratory objectives are:

Document: SAP SOMNUS

Template No.: RWI\_TP\_BIOS0013 Revision 2


1.0


Reference: RWI WI BIOS0015



- 1. Identify the proportion of patients with narcolepsy (Type 1 and Type 2) diagnosed and managed in public hospitals in Spain.
- 2. Evaluate and describe the diagnosis and treatment management of patients with narcolepsy up to one year before diagnosis (this objective will be assessed through medical chart review).
- 3. Describe utilization of health care resources associated with narcolepsy patients in Spain, before diagnosis of narcolepsy

### 4. STUDY DESIGN

## 4.1 General Description

A multicenter, non-interventional, cross-sectional, study with retrospective medical chart review, conducted in public and private Spanish institutions which has been designed to describe the management of narcolepsy in adults' patients in real world practice in Spain.

The study will be conducted in a single visit, considering a fieldwork period of 16 months to enroll all patients. The patient will be enrolled in one of the two study cohorts according to the type of narcolepsy at the time of the visit and after patient informed consent is obtained:

• Cohort A: type 1 narcolepsy patients

• Cohort B: type 2 narcolepsy patients

Target population will be patients with confirmed diagnosis of narcolepsy defined by the International Classification of Sleep Disorders, Third Edition (ICDS-3), up to 7 years before study inclusion.

### **Determination of sample size**

Document: SAP SOMNUS


1.0

Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Oct2021



The main objective of this study is to describe treatment patterns of narcolepsy patients in Spain.

Since it is an exploratory analysis, the sample size (N) will be calculated based on statistical criteria, using the criterion of maximum indetermination, when the percentage is expected to be around 50%.

A sample of 196 evaluable patients is sufficient to estimate a population percentage of 50%, with a 95% confidence interval of  $\pm$  7 percentage units. In this way, the continuous variables will be estimated with an accuracy of 0.14 standard deviations (SD).

Considering that around 20% of patients will not have any evaluable data or will be not considered evaluable for the study purposes, the number of patients with narcolepsy to be included will be approximately 245 patients: 172 patients with type 1 narcolepsy and 73 patients with type 2 narcolepsy (a relation of 70%-30%).

### 4.2 Schedule of Events

The schedule of events can be found in Section 4.1 of the protocol.

# 4.3 Changes to Analysis from Protocol

No changes in analysis or definitions included in the final protocol have been considered.

### 5. PLANNED ANALYSES

### 5.1 Interim Analysis

No interim analyses are planned for this study.

## 5.2 Final Analysis

Template No.: RWI\_TP\_BIOS0013 Revision 2

All final, planned analyses identified in this SAP will be performed by IQVIA Real World (RW) Biostatistics following IQVIA SOPs. Final CSR will be performed using IQVIA template.

Document: SAP SOMNUS

Author:


Reference: RWI\_WI\_BIOS0015



### 6. ANALYSIS SETS

# 6.1 All Subjects Enrolled Set [ENR]

The all subjects enrolled (ENR) set will contain all subjects who provide informed consent for this study and fulfilling all inclusion and none of exclusion criteria.

### 6.1.1 Inclusion criteria

Subject eligibility is determined according to the following criteria prior to inclusion into the study:

- 1. Patient aged ≥18 years at the time of study inclusion
- 2. Patient with confirmed diagnosis of narcolepsy defined by the International Classification of Sleep Disorders, Third Edition (ICDS-3)
- 3. Patient with at least 1-year follow-up with data available at the participating site after initial narcolepsy diagnosis and before study inclusion.
- 4. Patients with data available at the participant site at least 1-year before first narcolepsy diagnosis
- 5. Patient capable to fulfill the study questionnaires.
- 6. In the opinion of the investigator, the subject is capable of understanding and complying with protocol requirements.
- 7. The subject or, when applicable, the subject's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.

### 6.1.2 Exclusion criteria

Any subject who meets any of the following criteria will not qualify for entry into the study:

- 1. Patient with any serious degenerative disease (Alzheimer, Parkinson or epilepsy) or psychiatric condition
- 2. Any other reason that, in the Investigator's opinion, makes the patient unsuitable to participate in this study.

Document: SAP S

SAP SOMNUS

Author:


1.0


Reference: RWI\_WI\_BIOS0015

E#--#-- D-4-- 450-40004

Template No.: RWI\_TP\_BIOS0013 Revision 2



3. Patient participating in a clinical trial (≤12 months\*)

\*Clinical trial participation could be cause of bias regarding healthcare resource use data collection.

Subjects should be included in the study only once.

Data erroneously collected from subjects for which written consent is not available, will not be included in or will be deleted from the database.

### 6.2 Safety Analysis Set [SAF]

The safety analysis set (SAF) will contain all enrolled patients who received at least one dose of narcolepsy treatments.

If there is any doubt whether a patient was treated or not, they will be assumed treated for the purposes of analysis.

# 7. GENERAL CONSIDERATIONS

Patients will attend a single visit where they will answer study questionnaires and some clinical variables will be collected from clinical records.

Data will be collected:

- **Retrospective Period:** patient should have at least 1 year of follow-up before narcolepsy diagnosis and must have been diagnosed of narcolepsy, having at least 1 year of follow-up before study visit.
- **Study visit:** Clinical and demographic data and PRO will be collected from the patient during the study visit, respectively.

Considering the study design, 3 periods of time will be considered:

• **Index Period** will be the period in which patient is diagnosed of narcolepsy.

Document: SAP SOMNUS
Author:


Reference: RWI\_WI\_BIOS0015

Effective Date: 15Oct2021

Template No.: RWI\_TP\_BIOS0013 Revision 2



- **Post-Index** will be the at least a 1-year period before study visit all patients must have for the collection of use of resources in the last year
- **Pre-Index period** will 12 months before diagnosis (for the exploratory objective)

#### 7.1 **Windowing Conventions**

No visit windowing will be performed for this study.

#### 7.2 **Collected Variables and Measures**

Only variables included in the CRF will be used in this analysis. To describe real-world management and treatment patterns in narcolepsy patients in Spain, periods of time will be considered.

#### 7.2.1 **Primary endpoint**

To achieve the primary objective of this study, describe the treatment patterns of narcolepsy, the following endpoints will be collected and analyzed:

- Percentage of use of treatments (pharmacological and non-pharmacological) (yes / no) in the study visit
  - Total narcolepsy population
    - Patients with Type 1 and Type 2 narcolepsy
- Use of different treatments (pharmacological and non-pharmacological) in the study visit
  - Total narcolepsy population
  - Stratified by the different subgroups
    - Patients with Type 1 and Type 2 narcolepsy
    - Patients treated and treatment-naïve patients

SAP SOMNUS Document:

Author:

Template No.: RWI\_TP\_BIOS0013 Revision 2


Reference: RWI WI BIOS0015



A description of non-pharmacological treatments (since diagnosis): Take short naps; Maintain
a regular sleep schedule; Avoid caffeine or alcohol before bed; Avoid smoking, especially at
night; Exercise daily; Avoid large, heavy meals right before bedtime; Other

Also, a description of percentage of use of each type of treatment in the study visit will be stratified by type of hospital (public or private centers).

## 7.2.2 Secondary endpoints

Below is detailed the secondary objectives of this study and all secondary endpoints that will be collected and analyzed to achieve them:

- Describe sociodemographic and clinical characteristics of patients with narcolepsy
  - Sociodemographic and clinical characteristics (general clinical history and narcolepsy characteristics) of patients with narcolepsy collected in the study visit will be presented stratified by treatment-naïve patients and treated patients. Comparisons between groups will be performed using a Chi-Square test for categorical variables and t-test or non-parametric test for continuous variables.
- To describe specialists involved in diagnosis of patients with narcolepsy
  - o The percentage of different specialists who diagnosed narcolepsy will be presented
- To describe diagnosis processes used in real-world as described in patients' medical records
  - The percentage of the different procedures or tests for the diagnosis of narcolepsy will be described: clinical history, (absence/presence of cataplexy, number of cataplexy attacks, number of sleep-onset REM periods (SOREMPs), absence/presence of apneas and /or Apnea-hypopnea index (AHI), ESS, PSG, MSLT and HLA haplotypes will be described.

Document:

SAP SOMNUS

Author:

Version Number: Version Date:

[19JAN2023]

1.0

Reference: RWI\_WI\_BIOS0015

Template No.: RWI\_TP\_BIOS0013 Revision 2



- Time since first symptoms to diagnosis and time from diagnosis to first treatment will be described.
- To evaluate and describe clinician assessments (effectiveness) of the used narcolepsy treatments in the study period:
  - Percentage of treatments in which information on scales used to measure treatment outcomes is available: ESS, MWT and SART at the study visit will be described and the relation with the treatment received.
- To estimate direct and indirect healthcare resources utilization use by narcolepsy patients in Spain, based on measures of healthcare resource utilization, and on reported work productivity loss the 12 months before study visit in terms:
  - Direct medical healthcare resources used by patients with narcolepsy will be described in terms of percentage of patients who used each direct healthcare resource in the las 12 months prior to study visit including previous treatments for narcolepsy, outpatient visits, clinical tests, emergency room/department visits, hospitalizations and complication associated to narcolepsy. Also, it will be described the number of each type of direct resources used by patient/year (assuming as zero when patients did not used it). To compute total cost, the following direct cost components will be summed for fees for visits to doctors, laboratory tests and imaging tests, outpatient visits, emergency room visits, inpatient stays, rehabilitation stays, and drug treatments related to MS. The monetary cost will not be calculated.
  - Indirect health resources in the last 7 days will be described through the WPAI questionnaire scores obtained for:

Document:

SAP SOMNUS

Template No.: RWI\_TP\_BIOS0013 Revision 2

Author:


1.0


Reference: RWI\_WI\_BIOS0015



- 1. Absenteeism (work time missed).
- 2. Presenteeism (impairment at work / reduced on-the-job effectiveness)
- 3. Work productivity loss (overall work impairment / absenteeism plus presenteeism)
- 4. Activity Impairment / disability.
- o Indirect health care due to occupational accidents motor vehicle accidents (MVAs) and near miss accidents (NMAs) will also be described, through the answer of the two following questions: Have you had a motor vehicle accident at work during the last years?", "Have you had a near-miss driving accident during the last year?
- To describe the Health-Related Quality of Life (HRQoL) of patients with narcolepsy in Spain:
  - The EQ-5D scores of patients with narcolepsy in Spain will be described according to the following dimensions
    - Mobility
    - Self-Care
    - Usual activities
    - Pain / Discomfort
    - Anxiety / Depression
    - EQ VAS
- To assess the perception of stigma in patients with narcolepsy in Spain:
  - To know the level of stigmatization of patients with narcolepsy the score in the SSCI-8 will be described.

• To describe treatment satisfaction of patients with narcolepsy in Spain

Document: SAP SOMNUS
Author:

Template No.: RWI\_TP\_BIOS0013 Revision 2


Reference: RWI\_WI\_BIOS0015



- TSQM-9 domains will be described, including convenience, effectiveness and global satisfaction.
- To describe burden of illness in terms of associated comorbidities and associated disorders
  - Percentages (%) of most prevalent comorbidities and other concomitant disorders associated with narcolepsy will be described.
  - O Charlson Comorbidity Index(25) (CCI), score is a method to estimate 10-year mortality based on a score from a range of 12 comorbidities, the comorbidity score ranges from 0 to a maximum of 24 points.
- To describe adverse reaction associated to narcolepsy treatments
  - Describe type of adverse events (AE) reported

# 7.2.3 Exploratory endpoints

- Identify the proportion of patients with narcolepsy (with and without cataplexy) diagnosed and managed in public hospitals in Spain
  - The percentage of total number of patients with narcolepsy attended in the participating site according to routine clinical practice with at least 12-months follow up after over total population under the hospital's circumscription.
  - New patients diagnosed with narcolepsy in the last year in the participating sites over total population under the hospital's circumscription.

Document:

SAP SOMNUS

Template No.: RWI\_TP\_BIOS0013 Revision 2

Author:


1.0


Reference: RWI\_WI\_BIOS0015



- Evaluate and describe the diagnosis and treatment management of patients with narcolepsy up to one year before diagnosis (if this information is not available in the medical charts, this objective will be assessed through a patient survey).
  - O Description (%) treatments received for narcolepsy in the last year before diagnosis will be described.
- Describe utilization of health care resources associated with narcolepsy patients in Spain, before diagnosis of narcolepsy
  - o Description (quantity and type) of healthcare resources associated with narcolepsy patients 12 months before being diagnosed for this condition.

    Other analysis

## 7.2.4

Different general linear models (GLM) for the continuous healthcare resources (number of visits, number of tests, number of hospitalizations,... the 12 months before study visit) will be estimated using continuous and/or categorical variables, with a p-value<0.1 at univariate level. Predictors such as age, gender, time since diagnosis, type of narcolepsy will be evaluated. According to the distribution of the dependent variable, logistic regression models will be considered according to the use or non-use of the resource.

In the same way, three models will be carried out to evaluate the predictive factors of QoL (EQ VAS), stigma (SSCI-8 score) and satisfaction (TSQM-9 global satisfaction score).

All those tables presented in section 18 of this document and that are stratified by type of narcolepsy will be analyzed in addition to type of narcolepsy by type of center (public or private). These tables will be included in an annex to the statistical report.

Document: SAP SOMNUS

Author:

Template No.: RWI\_TP\_BIOS0013 Revision 2


Reference: RWI WI BIOS0015



#### 7.3 **Software Version**

All analyses will be conducted using SAS Enterprise Guide 7.15 or higher.

#### 8. STATISTICAL CONSIDERATIONS

#### 8.1 **Statistical Tests and Confidence Intervals**

A two-sided 95% confidence interval will be considered as a default (alpha= 5%). To analyze statistically significant differences between qualitative variables included as the secondary objective sociodemographic and clinical characteristics of patients with narcolepsy (gender and ethnicity), Chi-Square test, while for quantitative variables included in the same objective (such as age) t-test or Mann-Whitney non-parametric test according to the distribution of data.

#### Adjustments for Covariates and Factors to be Included in Analyses 8.2

No covariates and factor will be used in the analyses.

#### 8.3 Missing data

Given the real-world nature and retrospective part of the study and the descriptive purposes of most of the objectives included, study variables will not be imputed.

Missing values and drop-outs will be counted in all description of variables, but no imputation will be considered in this study.

#### 8.4 **Examination of Subgroups**

The variables description (primary, secondary, and exploratory) will be divided by groups. The following subgroups will be assessed:

- Type of narcolepsy
  - Type 1 (NT1)
  - Type 2 (NT2)

Document:

SAP SOMNUS

Template No.: RWI\_TP\_BIOS0013 Revision 2

Author:


1.0

Reference: RWI WI BIOS0015



- Previous treatment (secondary objective 1)
  - Treated
  - Untreated (naïve): Patients who have not received any pharmacological treatment from diagnosis to study visit.

### 8.5 Derived variables

Some variables will be calculated to be analyzed:

- Patients untreated (naïve): Percentage of patients with narcolepsy who are not with any pharmacological treatment from diagnosis to study visit.
- Patients treated: Percentage of patients with narcolepsy whose are with any pharmacological treatment.

### 9. OUTPUT PRESENTATIONS

Appendix 1 shows conventions for presentation of data in outputs.

# 10. DISPOSITION AND WITHDRAWALS

All subjects who provide informed consent will be accounted for in this study.

Subject disposition, withdrawals, and protocol violations (as defined in section 6.3), including inclusion and exclusion criteria will be presented for all enrolled patients.

### 11. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Demographic data and other baseline characteristics will be presented for all subjects enrolled (ENR). The following demographic and other baseline characteristics will be reported for this study:

• Age at the time of the visit

Template No.: RWI\_TP\_BIOS0013 Revision 2

Document: SAP SOMNUS
Author:


Reference: RWI\_WI\_BIOS0015



- Gender
- Ethnicity
- Educational level ongoing or completed level of education
- Occupational status and occupation
- Civil status
- Living conditions
- Height at treatment start (or last available before treatment initiation)
- Weight at treatment start (or last available before treatment initiation)
- BMI
- Blood pressure
- Smoking status
- Alcohol intake
- Exercise status
- Family history of narcolepsy in first or second-degree relatives

### 12. MEDICAL HISTORY

Medical History information will be presented for the ENR. This information will be collected from the CRF corresponding sections.

### 13. CONCOMITANT ILLNESSES

Concomitant illnesses will be presented for the ENR.

Comorbidities and other narcolepsy-associated disorders reported during the study period will be collected from comorbidities section and other narcolepsy associated disorders and concomitant treatment experienced by the patient during the study period page of the CRF.

Document: SAP SOMNUS

Author:

Template No.: RWI\_TP\_BIOS0013 Revision 2


1.0


Reference: RWI\_WI\_BIOS0015

### 14. MEDICATIONS

Medications will be presented for the ENR. It will include all treatments received the 12 months before the diagnosis of narcolepsy and also 12 months before study visit.

There will be six groups of medications according to the study groups:

- Stimulants
- Wakefulness-promoting agents
- Sodium Oxybate
- Antidepressants
- Benzodiazepines
- Other psychotropic agents

# 15. PATIENT REPORTED OUTCOMES (PRO)

At the study visit, patients several PROS will completed:

- Work Productivity and Activity Impairment Questionnaire General (WPAI-GH)
- EQ-5D Questionnaire
- Stigma Scale for Chronic Illness 8-item version (SSCI-8)
- Treatment Satisfaction Questionnaire for Medication (TSQM-9)

### 15.1 WPAI-GH

Work Productivity and Activity Impairment Questionnaire General (WPAI-GH) will be used to estimated indirect health resources used. It will be obtained for:

- Absenteeism (work time missed): Q2/(Q2+Q4) x100
- o Presenteeism (impairment at work / reduced on-the-job effectiveness): Q5/10 x100


1.0

Document: SAP SOMNUS


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Oct2021



- O Work productivity loss (overall work impairment / absenteeism plus presenteeism): Q2/(Q2+Q4)+[(1-(Q2/(Q2+Q4)))x(Q5/10)]x100
- o Activity Impairment / disability: Q6/10 x100

Information will be described as mean and standard deviation, median and interquartile range, minimum and maximum values. Valid and missing values will be also included.

### 15.2 EQ-5D

Quality of Life (QoL) will be assess using EQ-5D questionary. The information will be described according to the following dimensions:

- Mobility
- Self-Care
- Usual activities
- o Pain / Discomfort
- Anxiety / Depression

Information will be described as number and percentage of patients with problems in each dimension. Valid and missing values will be also included.

### 15.3 SSCI-8

Regarding Stigma Scale for Chronic Illness 8-item version (SSCI-8), data will be described as mean and standard deviation, median and interquartile range, minimum and maximum values. Valid and missing values will be also included. SSCI-8 raw score will be calculated summing individual items. Stigma prevalence will be calculated (total score>8). It will be describing a frequency and percentage.

### 15.4 TSQM-9

Treatment Satisfaction Questionnaire for Medication (TSQM-9) domains will be described, including convenience, effectiveness, and global satisfaction.

Document: SAP SOMNUS

Author:

Template No.: RWI\_TP\_BIOS0013 Revision 2


Reference: RWI\_WI\_BIOS0015



EFFECTIVENESS ([(Item 1 + Item 2 + Item 3) - 3] divided by 18) \* 100 If one item is missing ([(Sum(Item 1? + Item 2? + Item 3?)) - 2] divided by 12) \* 100

CONVENIENCE ([(Item 4 + Item 5 + Item 6) - 3] divided by 18) \* 100 If one item is missing ([(Sum(Item 4? + Item 5? + Item 6?)) - 2] divided by 12) \* 100

GLOBAL SATISFACTION ([(Item 7 + Item8 + Item 9) - 3] divided by 14) \* 100 If either Item 7 or 8 is missing ([((Item7? + Item8? + Item 9)) - 2] divided by 10) \* 100 If Item 9 is missing ([((Item7 + Item9)) - 2] divided by 8) \* 100

Data will be reported as mean and standard deviation, median and interquartile range, minimum and maximum values. Valid and missing values will be also included.

# 16. SAFETY OUTCOMES

All outputs for safety outcomes will be based on the Safety Analysis Set. AEs were classified according to the Medical Dictionary for Regulatory Activities (MedDRA). A description of AEs (related and not related to Takeda product) will be done, according to SOC and PT.

Document: SAP SOMNUS


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Oct2021

Author:


1.0



#### 17. REFERENCES

Statistical Analysis Plan

- Sarkanen T, Alakuijala A, Partinen M. Ullanlinna Narcolepsy Scale in diagnosis of narcolepsy. Sleep. 1. 2019;42(3):zsy238.
- Ohayon MM, Priest RG, Zulley J, Smirne S, Paiva T. Prevalence of narcolepsy symptomatology and diagnosis in the European general population. Neurology. 2002;58(12):1826-33.
- Ohayon M, Priest R, Zulley J, Smirne S, Paiva T. Prevalence of narcolepsy symptomatology and diagnosis in 3. the European general population. Neurology. 2002;58(12):1826-33.
- Morrish E, King MA, Smith IE, Shneerson JM. Factors associated with a delay in the diagnosis of narcolepsy. Sleep medicine. 2004;5(1):37-41.
- Frauscher B, Ehrmann L, Mitterling T, Gabelia D, Gschliesser V, Brandauer E, et al. Delayed diagnosis, range of severity, and multiple sleep comorbidities: a clinical and polysomnographic analysis of 100 patients of the innsbruck narcolepsy cohort. Journal of clinical sleep medicine: JCSM: official publication of the American Academy of Sleep Medicine. 2013;9(8):805-12.
- Kornum BR, Knudsen S, Ollila HM, Pizza F, Jennum PJ, Dauvilliers Y, et al. Narcolepsy. Nature reviews 6. Disease primers. 2017;3:16100.
- Dunne L, Patel P, Maschauer EL, Morrison I, Riha RL. Misdiagnosis of narcolepsy. Sleep & breathing = Schlaf 7. & Atmung. 2016;20(4):1277-84.
- 8. Barateau L, Dauvilliers Y. Recent advances in treatment for narcolepsy. Therapeutic advances in neurological disorders. 2019;12:1756286419875622.
- de Biase S, Nilo A, Gigli GL, Valente M. Investigational therapies for the treatment of narcolepsy. Expert opinion on investigational drugs. 2017;26(8):953-63.
- Dauvilliers Y, Arnulf I, Mignot E. Narcolepsy with cataplexy. Lancet (London, England). 2007;369(9560):499-10. 511.
- Bhattarai J, Sumerall S. Current and Future Treatment Options for Narcolepsy: A Review. Sleep science (Sao 11. Paulo, Brazil). 2017;10(1):19-27.
- Cohen A, Mandrekar J, Louis EKS, Silber MH, Kotagal S. Comorbidities in a community sample of narcolepsy. 12. Sleep medicine. 2018;43:14-8.
- Thorpy MJ, Hiller G. The Medical and Economic Burden of Narcolepsy: Implications for Managed Care. 13. American health & drug benefits. 2017;10(5):233-41.
- Emsellem HA, Thorpy MJ, Lammers GJ, Shapiro CM, Mayer G, Plazzi G, et al. Measures of functional outcomes, work productivity, and quality of life from a randomized, phase 3 study of solriamfetol in participants with narcolepsy. Sleep medicine. 2020;67:128-36.
- Kok SW, Overeem S, Visscher TL, Lammers GJ, Seidell JC, Pijl H, et al. Hypocretin deficiency in narcoleptic 15. humans is associated with abdominal obesity. Obesity research. 2003;11(9):1147-54.
- Dauvilliers Y, Jaussent I, Krams B, Scholz S, Lado S, Levy P, et al. Non-dipping blood pressure profile in narcolepsy with cataplexy. PloS one. 2012;7(6):e38977.
- Plazzi G, Ferri R, Antelmi E, Bayard S, Franceschini C, Cosentino FI, et al. Restless legs syndrome is frequent 17. in narcolepsy with cataplexy patients. Sleep. 2010;33(5):689-94.
- Jennum P, Ibsen R, Petersen ER, Knudsen S, Kjellberg J. Health, social, and economic consequences of narcolepsy: a controlled national study evaluating the societal effect on patients and their partners. Sleep medicine. 2012;13(8):1086-93.
- Flores NM, Villa KF, Black J, Chervin RD, Witt EA. The Humanistic and Economic Burden of Narcolepsy. Journal of clinical sleep medicine: JCSM: official publication of the American Academy of Sleep Medicine. 2016;12(3):401-7.

Document: SAP SOMNUS

Template No.: RWI\_TP\_BIOS0013 Revision 2


Reference: RWI WI BIOS0015

Effective Date: 15Oct2021



- 20. Daniels E, King MA, Smith IE, Shneerson JM. Health-related quality of life in narcolepsy. Journal of sleep research. 2001;10(1):75-81.
- 21. Reilly MC, Zbrozek AS, Dukes EM. The validity and reproducibility of a work productivity and activity impairment instrument. Pharmacoeconomics. 1993;4(5):353-65.
- 22. Herdman, M., Gudex, C., Lloyd, A. et al. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res 20, 1727–1736 (2011). https://doi.org/10.1007/s11136-011-9903-x
- 23. Molina Y, Choi SW, Cella D, Rao D. The stigma scale for chronic illnesses 8-item version (SSCI-8): development, validation and use across neurological conditions. International journal of behavioral medicine. 2013;20(3):450-60.
- 24. Sweileh WM, Ihbesheh MS, Jarar IS, Taha ASA, Sawalha AF, Sa'ed HZ, et al. Self-reported medication adherence and treatment satisfaction in patients with epilepsy. Epilepsy & Behavior. 2011;21(3):301-5.
- 25. Quan H, Li B, Couris CM, Fushimi K, Graham P, Hider P, et al. Updating and validating the Charlson comorbidity index and score for risk adjustment in hospital discharge abstracts using data from 6 countries. American journal of epidemiology. 2011;173(6):676-82.

Document: SAP SOMNUS


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015

Effective Date: 15Oct2021

Author:


1.0



### 18. APPENDIX 1. PROGRAMMING CONVENTIONS FOR OUTPUTS

Total column will include description of total evaluable sample (ENR). Main analysis will be presented stratified by subgroups group according to objectives.

### 18.1 Inclusion-exclusion criteria

Table 1. Patients' validation criteria

| PATIENT INCLUSION CRITERIA, n (%) | Total |
|---|---|
| 1. Patient aged ≥18 years at the time of study inclusion | |
| 2. Patient with confirmed diagnosis of narcolepsy defined by the International | |
| Classification of Sleep Disorders, Third Edition (ICDS-3) | |
| 3. Patient with at least 1-year follow-up with data available at the participating site | |
| after initial narcolepsy diagnosis and before study inclusion. | |
| 4. Patients with data available at the participant site at least 1-year before narcolepsy | |
| diagnosis | |
| 5. Patient capable to <b>fulfill</b> the study questionnaires. | |
| 6. In the opinion of the investigator, the subject is capable of understanding and | |
| complying with protocol requirements. | |
| 7. The subject or, when applicable, the subject's legally acceptable representative signs | |
| and dates a written, informed consent form and any required privacy authorization prior | |
| to the initiation of any study procedures | |
| PATIENT EXCLUSION CRITERIA, n (%) | |
| 1.Patient with any serious degenerative disease (Alzheimer, Parkinson or epilepsy) or psychiatric condition | |
| 2. Any other reason that, in the Investigator's opinion, makes the patient unsuitable to | |
| participate in this study | |
| 3.Patient participating in a clinical trial (≤12 months) | |
| Total patients enrolled (ENR) | |
| Narcolepsy Type 1 (NT1) | |
| Narcolepsy Type 2 (NT2) | |
| Not Classified* | |

<sup>\*</sup>These patients will be excluded from the analysis. If there are enough cases, the characteristics of these patients will be described separately.

Document: SAP SOMNUS


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



# 18.2 Demographic and baseline characteristics

Table 2. Patients' sociodemographic and baseline characteristics

| | | NT1 | NT2 | Total | p-value |
|---|---|---|---|---|---|
| Age at the time of the visit, | Mean (SD) | | | | |
| years | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Gender, n (%) | Male | | | | |
| | Female | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Ethnicity, n (%) | Caucasian | | | | |
| | Hispanic | | | | |
| | African | | | | |
| | Asian / Oriental | | | | |
| | Other | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Educational level ongoing or | Without studies | | | | |
| completed level of education, n (%) | Primary Studies | | | | |
| (70) | Secondary Studies | | | | |
| | University Studies | | | | |
| | Other Superior Studies | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Occupational status and | Student | | | | |
| occupation, n (%) | Employed | | | | |
| | Self-employed | | | | |
| | Employed but on sick leave due to the study disease | | | | |

Document: SAP SOMNUS


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



| | | NT1 | NT2 | Total | p-value |
|---|---|---|---|---|---|
| | Permanent incapacity to work due to the study disease | | | | |
| | Permanent incapacity to work due to other reasons | | | | |
| | Unemployed | | | | |
| | Retired | | | | |
| | Domestic work | | | | |
| | Other | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Civil status, n (%) | Married/with partner | | | | |
| | Divorced/separated | | | | |
| | Unmarried | | | | |
| | Widow/er | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Living conditions, n (%) | Alone | | | | |
| | Wife/Husband and /or sons | | | | |
| | Family Caregivers | | | | |
| | Other Caregivers | | | | |
| | Valid N | | | | |
| | N missing | | | | |

Table 3. Patients' physical examination at study visit

| | | NT1 | NT2 | Total | p-value |
|---|---|---|---|---|---|
| Height at treatment start or last available | Mean (SD) | | | | |
| before treatment initiation, cm | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Weight at treatment start or last | Mean (SD) | | | | |
| available before treatment initiation, kg | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |

Document: SAP SOMNUS


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



| | | NT1 | NT2 | Total | p-value |
|---|---|---|---|---|---|
| | Valid N | | | | |
| | N missing | | | | |
| BMI, kg/m <sup>2</sup> | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Blood pressure (systolic), mmHg | Mean (SD) | | | | |
| | Median (Q1-Q3) | 121 | | | |
| | Min-Max | 30/13 | | | |
| | Valid N | a, 0 | | | |
| | N missing | | | | |
| Blood pressure (diastolic), mmHg | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Smoking status, n(%) | Current Smoker | | | | |
| | Ex-Smoker | | | | |
| | Non-Smoker | | | | |
| , | Valid N | | | | |
| | N missing | | | | |
| Alcohol intake, n(%) | Never | | | | |
| | Once or less per month | | | | |
| | 2-4 times per month | | | | |
| | 2-3 times per week | | | | |
| | 4 or more times per week | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Exercise status, n(%) | Never | | | | |
| | Regular (1 - 3times/week) | | | | |
| | Frequently (4 - 7 times /week) | | | | |

Document: SAP SOMNUS


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



| | | NT1 | NT2 | Total | p-value |
|---|---|---|---|---|---|
| | Always (7 or more times/week) | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Family history of narcolepsy in first- or | No | | | | |
| second-degree relatives, n (%) | Yes | | | | |
| | First-degree relatives | | | | |
| | Second-degree relatives | | | | |
| | Valid N | | | | |
| | N missing | 121 | | | |

# 18.3 Diagnosis of narcolepsy

Table 4. Specialists involved in diagnosis of patients with narcolepsy (secondary objective 2)

| | NT1 | NT2 | Total | p-value |
|-----------------------------|-----|-----|-------|---------|
| General Practitioner, n (%) | 0, | | | |
| Specialist, n (%) | | | | |
| Specialist 1 | | | | |
| Specialist 2 | | | | |
| Specialist 3 | | | | |
| Specialist | | | | |
| Valid N | | | | |
| N missing | | | | |

Table 5. Time since first symptoms to diagnosis, time from diagnosis to first treatment and symptoms at diagnosis (secondary objective 3)

| | NT1 | NT2 | Total | p-value |
|-----------|-----|-----|-------|---------|
| Mean (SD) | | | | |

Document: SAP SOMNUS


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



| | | NT1 | NT2 | Total | p-value |
|---|---|---|---|---|---|
| Time since first symptoms to | Median (Q1-Q3) | | | | |
| diagnosis | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Another disease related to narcolepsy | No | | | | |
| of psychiatric disorders prior to | Yes | | | | |
| diagnosis of narcolepsy, n (%) | Type 1 | | | | |
| | Type 2 | | | | |
| | Specialist 1 | | | | |
| | Specialist 2 | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Time from diagnosis to first | Mean (SD) | | | | |
| pharmacological treatment | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Time from diagnosis to study visit | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Symptoms at diagnosis, n (%) | None | | | | |
| | Excessive daytime sleepiness (EDS) | | | | |
| | Cataplexy | | | | |
| | Hallucinations upon awakening or going to | | | | |
| | Sleep paralysis | | | | |
| | Disturbed night-time sleep | | | | |
| | Others | | | | |
| | Outers | | | | |

Document: SAP SOMNUS


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



| | | NT1 | NT2 | Total | p-value |
|---|---|---|---|---|---|
| | Valid N | | | | |
| | N missing | | | | |
| Number of cataplexy attacks per week before diagnosis | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |

Table 6. Procedures or tests for the diagnosis of narcolepsy (secondary objective 3)

| | | NTI | NT2 | Total | p-value |
|---|---|---|---|---|---|
| Clinical history, n (%) | | 5 | | | |
| Clinical Assessment: Epwo | rth sleepiness scale (ESS), n(%) | 3 | | | |
| | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| ESS score | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Neurological Assessment, r | 1 (%) | | | | |
| Polysomnogram (P | SG), n (%) | | | | |
| REM sleep latency | in nocturnal PSG, n (%) | | | | |
| Multiple sleep latency test ( | (MSLT), n (%) | | | | |
| | Mean (SD) | | | | |
| Number of sleep-onset | Median (Q1-Q3) | | | | |
| REM periods | Min-Max | | | | |
| (SOREMPs) | Valid N | | | | |
| | N missing | | | | |
| | Mean (SD) | | | | |
| Mean sleep latency (min) | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |

Document: SAP SOMNUS

Author:


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



| | | NT1 | NT2 | Total | p-value |
|---|---|---|---|---|---|
| Apnea-hypopnea index (A | .HI), n (%) | | | | |
| | 5-14.9 | | | | |
| | 15-29.9 | | | | |
| Electroencephalogical Electrooculography Electromyography Recordings of resp Recordings of airfl Pulse oximetry Electrocardiograph Other | >30 | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Other procedures, n (%) | | | | | |
| Electroencephalog | graphy (EEG | | | | |
| Electrooculograph | y | | | | |
| Electromyography | ī | | ) | | |
| Recordings of res | piratorymovements in your chest and tummy | 0, | | | |
| Recordings of airf | low through your mouth and nose | \$ | | | |
| Pulse oximetry | : 2 | | | | |
| Electrocardiograpl | hy (ECG) | | | | |
| Other | 20 | | | | |
| HLA typing, n (%) | W, | | | | |
| HLA DQB * 0602 | c <sub>O</sub> , | | | | |
| QB1*0304 | | | | | |
| Other at diagnosis | 100 | | | | |
| Hypocretin-1 CSF or Orex | xin, n (%) | | | | |
| | Low ( $<$ or =110 pg/mL), which is | | | | |
| | indicative of type 1 narcolepsy Intermediate (ranges between 111-200 | | | | |
| Levels in pg(mL al | pg/mL) | | | | |
| diagnosis, n (%) | Normal (>200 pg/mL) | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| | Low (< or =110 pg/mL), which is | | | | |
| | indicative of type 1 narcolepsy Intermediate (ranges between 111-200 | | | | |
| Levels at study visit, n (%) | pg/mL) | | | | |
| | Normal (>200 pg/mL) | | | | |
| | Valid N | | | | |
| | N missing | | | | |

Document: SAP SOMNUS


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



| | NT1 | NT2 | Total | p-value |
|-----------|-----|-----|-------|---------|
| Valid N | | | | |
| N missing | | | | |

### 18.4 Comorbidities

Table 7. Most prevalent comorbidities and other concomitant disorders associated with narcolepsy (present during the study period) (secondary objective 10)

| | | NT1 | NT2 | Total | p-value |
|---|---|---|---|---|---|
| Comorbidities, n (%) | No | | | | |
| | Yes | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Type of comorbidities, n | Depression | | | | |
| (%) | On going at study visit | | | | |
| | Bipolar disorder | | | | |
| | Anxiety disorder | | | | |
| | Generalized anxiety disorder | | | | |
| | Post-traumatic stress disorder | | | | |
| | Social anxiety disorder | | | | |
| | Panic disorder | | | | |
| | Phobia disorder | | | | |
| | Obsessive compulsive disorder | | | | |
| | Diagnosis of attention deficit hyperactivity disorder (ADHD) | | | | |
| | Obesity | | | | |
| | Endocrine Disorders | | | | |
| | Myocardial infarction | | | | |
| | Urinary Incontinence | | | | |
| | Congestive heart failure (CHF) | | | | |
| | Peripheral vascular disease | | | | |

Document: SAP SOMNUS


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015


| | | NT1 | NT2 | Total | p-value |
|---|---|---|---|---|---|
| | Cardiovascular accident or transient ischemic attack (TIA) | | | | |
| | Dementia (This was an exclusion criteria) | | | | |
| | Chronic obstructive pulmonary disease (COPD) | | | | |
| | Connective tissue disease | | | | |
| | Peptic ulcer disease | | | | |
| | Liver Disease | | | | |
| | Mild | | | | |
| | Moderate to severe | | | | |
| | Diabetes Mellitus | 11/ | | | |
| | None or diet controlled | 2/ | | | |
| | Uncomplicated | | | | |
| | End-organ damage | | | | |
| | Hemiplegia | | | | |
| | Moderate to severe chronic kidney disease (CKD) | | | | |
| | Solid tumor | | | | |
| | Localized | | | | |
| | Metastatic | | | | |
| | Leukemia | | | | |
| | Lymphoma | | | | |
| | AIDS | | | | |
| | Others | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| Charlson comorbidity index | Min-Max | | | | |
| IIIUCX | Valid N | | | | |
| | N missing | | | | |

Document: SAP SOMNUS


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



Table 8. Treatment for comorbidities and other concomitant disorders associated with narcolepsy (during the study period)

| | | NT1 | NT2 | Total | p-value |
|---|---|---|---|---|---|
| Treatment for | Depression | | | | |
| comorbidities and concomitant disorders, n | Stimulants | | | | |
| (%) | Wakefulness- Promoting Agents | | | | |
| | Sodium Oxybate | | | | |
| | Gammahydroxybutyrate (GHB) | | | | |
| | Antidepressants | | | | |
| | Benzodiazepines | | 117 | | |
| | Other | C | | | |
| | Bipolar disorder | 50 | | | |
| | Stimulants | 0 | | | |
| | Wakefulness- Promoting Agents | | | | |
| | Sodium Oxybate | | | | |
| | Gammahydroxybutyrate (GHB) | | | | |
| | Antidepressants | | | | |
| | Benzodiazepines | | | | |
| | Other | | | | |
| | Anxiety disorder | | | | |
| | Stimulants | | | | |
| | Wakefulness- Promoting Agents | | | | |
| | Sodium Oxybate | | | | |
| | Gammahydroxybutyrate (GHB) | | | | |
| | Antidepressants | | | | |
| | Benzodiazepines | | | | |
| | Other | | | | |
| | Generalized anxiety disorder | | | | |
| | Stimulants | | | | |
| | Wakefulness- Promoting Agents | | | | |
| | Sodium Oxybate | | | | |
| | Gammahydroxybutyrate (GHB) | | | | |

Document: SAP SOMNUS


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



| | NT1 | NT2 | Total | p-value |
|-------------------------------|-----|-----|-------|---------|
| Antidepressants | | | | |
| Benzodiazepines | | | | |
| Other | | | | |
| Generalized anxiety disorder | | | | |
| Stimulants | | | | |
| Wakefulness- Promoting Agents | | | | |
| Sodium Oxybate | | | | |
| Gammahydroxybutyrate (GHB) | | | | |
| Antidepressants | | 14 | | |
| Benzodiazepines | Č | | | |
| Other | ~® | | | |
| Panic disorder | 113 | | | |
| Stimulants | | | | |
| Wakefulness- Promoting Agents | | | | |
| Sodium Oxybate | | | | |
| Gammahydroxybutyrate (GHB) | | | | |
| Antidepressants | | | | |
| Benzodiazepines | | | | |
| Other | | | | |
| Phobia disorder | | | | |
| Stimulants | | | | |
| Wakefulness- Promoting Agents | | | | |
| Sodium Oxybate | | | | |
| Gammahydroxybutyrate (GHB) | | | | |
| Antidepressants | | | | |
| Benzodiazepines | | | | |
| Other | | | | |
| Obsessive compulsive disorder | | | | |
| Stimulants | | | | |
| Wakefulness- Promoting Agents | | | | |
| Sodium Oxybate | | | | |
| Gammahydroxybutyrate (GHB) | | | | |

Document: SAP SOMNUS


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



| | NT1 | NT2 | Total | p-value |
|---|---|---|---|---|
| Antidepressants | | | | |
| Benzodiazepines | | | | |
| Other | | | | |
| Diagnosis of attention deficit hyperactivity disorder (ADHD) | | | | |
| Stimulants | | | | |
| Wakefulness- Promoting Agents | | | | |
| Sodium Oxybate | | | | |
| Gammahydroxybutyrate (GHB) | | | | |
| Antidepressants | | 17 | | |
| Benzodiazepines | Ċ | | | |
| Other | CO | | | |
| Obesity | 100 | | | |
| Endocrine Disorders | | | | |
| Treatment 1 | | | | |
| Myocardial infarction | | | | |
| Treatment 1 | | | | |
| Urinary Incontinence | | | | |
| Treatment 1 | | | | |
| Congestive heart failure (CHF) | | | | |
| Treatment 1 | | | | |
| Peripheral vascular disease | | | | |
| Treatment 1 | | | | |
| Cardiovascular accident or transient ischemic attack (TIA) | | | | |
| Treatment 1 | | | | |
| Dementia (exclusion criteria) | | | | |
| Treatment 1 | | | | |
| Chronic obstructive pulmonary disease (COPD) | | | | |
| Treatment 1 | | | | |
| Connective tissue disease | | | | |

Document: SAP SOMNUS


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



| | | NT1 | NT2 | Total | p-value |
|---|---|---|---|---|---|
| Per | ptic ulcer disease | | | | |
| | Treatment 1 | | | | |
| Liv | ver Disease | | | | |
| | Treatment 1 | | | | |
| Dia | abetes Mellitus | | | | |
| | Treatment 1 | | | | |
| Her | miplegia | | | | |
| | Treatment 1 | | | | |
| | oderate to severe chronic kidney ease (CKD) | | K | | |
| | Treatment 1 | Ó | | | |
| Sol | lid tumor | S | | | |
| | Treatment 1 | 7, | | | |
| Lei | ukemia | | | | |
| | Treatment 1 | | | | |
| Lyı | mphoma | | | | |
| | Treatment 1 | | | | |
| AII | DS | | | | |
| | Treatment 1 | | | | |
| Oth | hers | | | | |
| | Treatment 1 | | | | |
| Val | lid N | | | | |
| Nr | missing | | | | |

Table 9. Most prevalent comorbidities and other concomitant disorders associated with narcolepsy (on going at study visit) (secondary objective 10)

| | | NT1 | NT2 | Total | p-value |
|----------------------|-----------|-----|-----|-------|---------|
| Comorbidities, n (%) | No | | | | |
| | Yes | | | | |
| | Valid N | | | | |
| | N missing | | | | |

Document: SAP SOMNUS


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



| | | NT1 | NT2 | Total | p-value |
|---|---|---|---|---|---|
| Type of comorbidities, n (%) | Depression | | | | |
| | Bipolar disorder | | | | |
| | Anxiety disorder | | | | |
| | Generalized anxiety disorder | | | | |
| | Post-traumatic stress disorder | | | | |
| | Social anxiety disorder | | | | |
| | Panic disorder | | | | |
| | Phobia disorder | | | | |
| | Obsessive compulsive disorder | 101 | | | |
| | Diagnosis of attention deficit hyperactivity disorder (ADHD) | 2013 | | | |
| | Obesity | | | | |
| | Endocrine Disorders | | | | |
| | Myocardial infarction | | | | |
| | Urinary Incontinence | | | | |
| | Congestive heart failure (CHF) | | | | |
| | Peripheral vascular disease | | | | |
| | Cardiovascular accident or transient ischemic attack TIA | | | | |
| | Dementia exclusion criteria | | | | |
| | Chronic obstructive pulmonary disease (COPD) | | | | |
| | Connective tissue disease | | | | |
| | Peptic ulcer disease | | | | |
| | Liver Disease | | | | |
| | Mild | | | | |
| | Moderate to sever | | | | |
| | Diabetes Mellitus | | | | |
| | None or diet controlled | | | | |
| | Uncomplicated | | | | |
| | End-organ damage | | | | |
| | Hemiplegia | | | | |
| | Moderate to severe chronic kidney disease (CKD) | | | | |

Document: SAP SOMNUS


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



| | | NT1 | NT2 | Total | p-value |
|----------------------------|----------------|------|-----|-------|---------|
| | Solid tumor | | | | |
| | Localized | | | | |
| | Metastatic | | | | |
| | Leukemia | | | | |
| | Lymphoma | | | | |
| | AIDS | | | | |
| | Others | | | | |
| | Valid N | | | | |
| | N missing | 121 | | | |
| | Mean (SD) | 1012 | | | |
| | Median (Q1-Q3) | 0. | | | |
| Charlson comorbidity index | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |

#### 18.5 **Treatment patterns**

Type of previous pharmacological treatment (treatments received in the 12 months Table 10. prior to diagnosis) according to type of narcolepsy (exploratory objective 2)

| | × · | NT1 | NT2 | Total | p-value |
|---|---|---|---|---|---|
| Treatment, n (%) | No | | | | |
| | Yes | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Type of treatment, n (%) | Stimulants | | | | |
| | Wakefulness-Promoting Agents | | | | |
| | Modafinil | | | | |
| | Pitolisant | | | | |
| | Solriamfetol | | | | |
| | Other | | | | |
| | Sodium Oxybate | | | | |

Document: SAP SOMNUS

Author: Version Number:


1.0

Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



| | NT1 | NT2 | Total | p-value |
|---------------------------|-----|-----|-------|---------|
| Antidepressants | | | | |
| Benzodiazepines | | | | |
| Other psychotropic agents | | | | |
| Valid N | | | | |
| N missing | | | | |

Table 11. Type of pharmacological treatment (1<sup>st</sup> treatment after diagnosis) according to type of narcolepsy (primary objective)

| | | NTI | NT2 | Total | p-value |
|---|---|---|---|---|---|
| 1st Treatment, n (%) | No | 0, | | | |
| | Yes | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Type of treatment, n (%) | Stimulants - monotherapy | | | | |
| | Wakefulness-Promoting Agents -<br>monotherapy | | | | |
| | Modafinil | | | | |
| | Pitolisant | | | | |
| | Solriamfetol | | | | |
| | Other | | | | |
| | Sodium Oxybate - monotherapy | | | | |
| | Antidepressants - monotherapy | | | | |
| | Benzodiazepines - monotherapy | | | | |
| | Other psychotropic agents - monotherapy | | | | |
| | Combinations (all combination to be described) | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Duration (in months) of first treatment | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |

Document: SAP SOMNUS

Author:


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



| | NT1 | NT2 | Total | p-value |
|-----------|-----|-----|-------|---------|
| N missing | | | | |

Table 12. Type of pharmacological treatment (since diagnosis up to study visit) according to type of narcolepsy (primary objective)

| | | NT1 | NT2 | Total | p-value |
|---|---|---|---|---|---|
| Treatment, n (%) | No | | | | |
| | Yes | 17 | | | |
| | Valid N | OLLI | ) | | |
| | N missing | .0 | | | |
| Type of treatment, n (%) | Stimulants | | | | |
| | Wakefulness-Promoting Agents | | | | |
| | Modafinil | | | | |
| | Pitolisant | | | | |
| | Solriamfetol | | | | |
| | Other | | | | |
| | Sodium Oxybate | | | | |
| | Antidepressants | | | | |
| | Benzodiazepines | | | | |
| | Other psychotropic agents | | | | |
| | Combinations (modafenil, pitolisant, sodium Oxybate, solriamfetol)* | | | | |
| | Valid N | | | | |
| | N missing | | | | |

<sup>\*</sup> how these treatments combined with other treatments, independently of the line of treatment

Table 13. Type of non-pharmacological treatment since diagnosis according to type of narcolepsy (primary objective)

| | NT1 | NT2 | Total | p-value |
|----|-----|-----|-------|---------|
| No | | | | |

Document: SAP SOMNUS

Author:


Reference: RWI\_WI\_BIOS0015

Template No.: RWI\_TP\_BIOS0013 Revision 2



| | | NT1 | NT2 | Total | p-value |
|---|---|---|---|---|---|
| | Yes | | | | |
| Non-pharmacological treatment, n (%) | Valid N | | | | |
| treatment, if (70) | N missing | | | | |
| Type, n (%) | Take short naps | | | | |
| | Maintain a regular sleep schedule | | | | |
| | Avoid caffeine or alcohol before bedtime | | | | |
| | Avoid smoking, especially at night | | | | |
| | Exercise daily | | | | |
| | Avoid large, heavy meals right before bedtime | | | | |
| | Other | 4 | | | |
| | Valid N | 0, | | | |
| | N missing | , | | | |

Table 14. Type of non-pharmacological treatment since diagnosis according to treated or untreated patients (primary objective)

| | c <sub>O</sub> t | Naïve | Treated | Total | p-value |
|---|---|---|---|---|---|
| Non-pharmacological | No | | | | |
| treatment, n (%) | Yes | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Type, n (%) | Take short naps | | | | |
| | Maintain a regular sleep schedule | | | | |
| | Avoid caffeine or alcohol before bedtime | | | | |
| | Avoid smoking, especially at night | | | | |
| | Exercise daily | | | | |
| | Avoid large, heavy meals right before bedtime | | | | |
| | Other | | | | |
| | Valid N | | | | |
| | N missing | | | · | |

Document: SAP SOMNUS


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



Table 15. Type of pharmacological treatment (at study visit) according to type of narcolepsy (primary objective)

| | | NT1 | NT2 | Total | p-value |
|---|---|---|---|---|---|
| Treatment, n (%) | No | | | | |
| | Yes | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Type of treatment, n (%) | Stimulants | | | | |
| | Wakefulness-Promoting Agents | | | | |
| | Modafinil | 417 | | | |
| | Pitolisant | 0, | | | |
| | Solriamfetol | | | | |
| | Other | | | | |
| | Sodium Oxybate | | | | |
| | Antidepressants | | | | |
| | Benzodiazepines | | | | |
| | Combinations (all combinations to be described) | | | | |
| | Other psychotropic agents | | | | |
| | Valid N | | | | |
| | N missing | | | | |

Table 16. Clinician assessment (effectiveness) of the used narcolepsy treatments in the study period since diagnosis (secondary objective 4)

| | | Stimulants | Wakefulness-<br>Promoting<br>Agents | Modafinil | Pitolisant | Solriamfetol | Sodium<br>oxybate | Antidepressants | Benzodiazepines |
|---|---|---|---|---|---|---|---|---|---|
| NT1 (total) | | | | | | | | | |
| Effectiveness of treatment by | None | | | | | | | | |
| Clinician<br>Assessment | Assessment with scales | | | | | | | | |
| , n (%) | SART | | | | | | | | |
| | MWT | | | | | | | | |
| | ESS | | | | | | | | |

Document:

SAP SOMNUS

Author:


Reference: RWI\_WI\_BIOS0015

Template No.: RWI\_TP\_BIOS0013 Revision 2



| | | Stimulants | Wakefulness-<br>Promoting<br>Agents | Modafinil | Pitolisant | Solriamfetol | Sodium<br>oxybate | Antidepressants | Benzodiazepines |
|---|---|---|---|---|---|---|---|---|---|
| | Cataplexy scales | | | | | | | | |
| | Other assessments | | | | | | | | |
| | Other 1 | | | | | | | | |
| | Other 2 | | | | | | | | |
| | Valid N* | | | | | | | | |
| | N missing | | | | | | | | |
| SART value | Mean (SD) | | | | | . \ | | | |
| | Median (Q1-Q3) | | | | | 7/3 | | | |
| | Min-Max | | | | ,50 | ) ` | | | |
| | Valid N* | | | | US | | | | |
| | N missing | | | :\? | , | | | | |
| MWT minutes | Mean (SD) | | | O.C. | | | | | |
| | Median (Q1-Q3) | | 2 | lu. | | | | | |
| | Min-Max | | COL | | | | | | |
| | Valid N* | | OU. | | | | | | |
| | N missing | 4 | (1) | | | | | | |
| ESS score | Mean (SD) | €0, | | | | | | | |
| | Median (Q1-Q3) | | | | | | | | |
| | Min-Max | | | | | | | | |
| | Valid N* | | | | | | | | |
| | N missing | | | | | | | | |
| Cataplexy scale score | Mean (SD) | | | | | | | | |
| scare score | Median (Q1-Q3) | | | | | | | | |
| | Min-Max | | | | | | | | |
| | Valid N* | | | | | | | | |
| | N missing | | | | | | | | |
| NT2 | | | | | | | | | |

Document: SAP SOMNUS


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



| | | Stimulants | Wakefulness-<br>Promoting<br>Agents | Modafinil | Pitolisant | Solriamfetol | Sodium<br>oxybate | Antidepressants | Benzodiazepines |
|---|---|---|---|---|---|---|---|---|---|
| Effectiveness of treatment by | None | | | | | | | | |
| Clinician<br>Assessment | Assessment with scales | | | | | | | | |
| , n (%) | SART | | | | | | | | |
| | MWT | | | | | | | | |
| | ESS | | | | | | | | |
| | Cataplexy scales | | | | | | | | |
| | Other assessments | | | | | | | | |
| | Other 1 | | | | | 17 | | | |
| | Other 2 | | | | | | | | |
| | Valid N* | | | | J50 | | | | |
| | N missing | | | . 0 | | | | | |
| SART value | Mean (SD) | | | 40/6 | | | | | |
| | Median (Q1-Q3) | | | Us. | | | | | |
| | Min-Max | | -07 | | | | | | |
| | Valid N* | | | | | | | | |
| | N missing | | 0/. | | | | | | |
| MWT minutes | Mean (SD) | 101 | | | | | | | |
| | Median (Q1-Q3) | ~ | | | | | | | |
| | Min-Max | | | | | | | | |
| | Valid N* | | | | | | | | |
| | N missing | | | | | | | | |
| ESS score | Mean (SD) | | | | | | | | |
| | Median (Q1-Q3) | | | | | | | | |
| | Min-Max | | | | | | | | |
| | Valid N* | | | | | | | | |
| | N missing | | | | | | | | |
| | Mean (SD) | | | | | | | | |

Document: SAP SOMNUS


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



| | | Stimulants | Wakefulness-<br>Promoting<br>Agents | Modafinil | Pitolisant | Solriamfetol | Sodium<br>oxybate | Antidepressants | Benzodiazepines |
|---|---|---|---|---|---|---|---|---|---|
| | Median (Q1-Q3) | | | | | | | | |
| Cataplexy | Min-Max | | | | | | | | |
| scale score | Valid N* | | | | | | | | |
| | N missing | | | | | | | | |

<sup>\*</sup>N valid correspond to total of treatments

#### 18.6 Direct and indirect healthcare resources utilization

# 18.6.1 Healthcare resources in the last 12 months prior to study visit

Table 17. Direct medical healthcare resources used by patients – treatments in the last year prior to study visit (secondary objective 5)

| | | NT1 | NT2 | Total | p-value |
|---|---|---|---|---|---|
| Treatment, n (%) | No | | | | |
| | Yes | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Type of treatment, n (%) | Stimulants | | | | |
| | Wakefulness-Promoting Agents | | | | |
| | Modafinil | | | | |
| | Pitolisant | | | | |
| | Solriamfetol | | | | |
| | Other | | | | |
| | Sodium Oxybate | | | | |
| | Antidepressants | | | | |
| | Benzodiazepines | | | | |
| | Other psychotropic agents | | | | |
| | Valid N | | | | |
| | N missing | | | | • |

Document: SAP SOMNUS


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



Direct medical healthcare resources used by patients - Outpatients visits in the last Table 18. year (secondary objective 5)

| | | NT1 | NT2 | Total | p-value |
|---|---|---|---|---|---|
| Routine monitoring visits, n (%) | No | | | | |
| | Yes | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Total number of routine monitoring visits | Mean (SD) | | | | |
| | Median (Q1-Q3) | | 4 | | |
| | Min-Max | | 13 | | |
| | Valid N | 0 | | | |
| | N missing | Se | | | |
| Specialists involved, n (%) | General Practitioner | | | | |
| | Specialist | ) | | | |
| | Neurologist | | | | |
| | Neurophysiologist | | | | |
| | Psychiatris | | | | |
| | Other | | | | |
| | Other 1 | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Number of visits to General Practitioner | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Number of visits to Neurologist | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |

Document: SAP SOMNUS

Author:


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



| | | NT1 | NT2 | Total | p-value |
|---|---|---|---|---|---|
| Number of visits to Neurophysiologist | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Number of visits to Psychiatrist | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | 121 | | |
| | N missing | ۵, | 112 | | |
| Number of visits to other specialist | Mean (SD) | 0, | | | |
| | Median (Q1-Q3) | 15 | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |

Table 19. Direct medical healthcare resources used by patients – Tests conducted in the last year (secondary objective 5)

| | 4.0 | NT1 | NT2 | Total | p-value |
|---|---|---|---|---|---|
| Tests, n (%) | No | | | | |
| | Yes | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Total number of tests | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Tests conducted, n (%) | Clinical history | | | | |
| | Presence of cataplexy | | | | |
| | Neurological Assessment | | | | |

Document: SAP SOMNUS


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



| | | NT1 | NT2 | Total | p-value |
|---|---|---|---|---|---|
| | Clinical Assessment | | | | |
| | Determination of Hypocretin-1 CSF or Orexin | | | | |
| | Apnea-hypopnea index (AHI) | | | | |
| | Number of sleep-onset REM periods (SOREMPs) | | | | |
| | Epworth Sleepiness Scale (ESS) score | | | | |
| | PSG | | | | |
| | MSLT | | | | |
| | Laboratory | \ | | | |
| | Other | | | | |
| | Other 1 | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Number of clinical histories | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Number of Presence of cataplexy | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Number of Neurological Assessment | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Number of Clinical Assessment | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |

Document: SAP SOMNUS


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



| | | NT1 | NT2 | Total | p-value |
|---|---|---|---|---|---|
| | Valid N | | | | |
| | N missing | | | | |
| Number of determinations of | Mean (SD) | | | | |
| Hypocretin-1 CSF or Orexin | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Number of Apnea-hypopnea index | Mean (SD) | | | | |
| (AHI) | Median (Q1-Q3) | 1 | | | |
| | Min-Max | 377 | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Number of sleep-onset REM periods | Mean (SD) | | | | |
| (SOREMPs) | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Number of Epworth Sleepiness | Mean (SD) | | | | |
| Scale (ESS) | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Number of PSG | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Number of MSLT | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |

Document: SAP SOMNUS


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



| | | NT1 | NT2 | Total | p-value |
|------------------------|----------------|------|-----|-------|---------|
| Number of laboratories | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Number of Other | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | 9013 | | | |

Table 20. Direct medical healthcare resources used by patients – Emergency visits in the last year (secondary objective 5)

| | . (O' | NT1 | NT2 | Total | p-value |
|---|---|---|---|---|---|
| Emergency visits, n (%) | No | | | | |
| | Yes | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Total number of emergency visits | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |

Table 21. Direct medical healthcare resources used by patients – Hospitalizations in the last year (secondary objective 5)

| | | NT1 | NT2 | Total | p-value |
|-------------------------|---------|-----|-----|-------|---------|
| Hospitalizations, n (%) | No | | | | |
| | Yes | | | | |
| | Valid N | | | | |

Document:

SAP SOMNUS

Author:


1.0

Reference: RWI\_WI\_BIOS0015

Template No.: RWI\_TP\_BIOS0013 Revision 2



| | | NT1 | NT2 | Total | p-value |
|---|---|---|---|---|---|
| | N missing | | | | |
| Total number of hospitalizations | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| Hospitalizations' duration (days) | Min-Max | | | | |
| | Valid N | | ď | 11,3 | |
| | N missing | | -61 | | |

Table 22. Direct medical healthcare resources used by patients – complications derived from narcolepsy in the last year (secondary objective 3)

| | orn't | NT1 | NT2 | Total | p-value |
|---|---|---|---|---|---|
| Complications, n (%) | No | | | | |
| | Yes | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Total number of complications | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Type of complications, n (%) | Obesity | | | | |
| | Interference with intimate relationships | | | | |
| | Fertility | | | | |
| | Physical harm: Attending to psychiatrist | | | | |
| | Work problems | | | | |
| | Others | | | | |
| | Other 1 | | | | |

Document: SAP SOMNUS


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



| | NT1 | NT2 | Total | p-value |
|-----------|-----|-----|-------|---------|
| Valid N | | | | |
| N missing | | | | |

Table 23. Indirect health resources - WPAI questionnaire scores (secondary objective 6)

| | | NT1 | NT2 | Total | p-value |
|---|---|---|---|---|---|
| Absenteeism | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | "13 | | |
| | N missing | | 0, | | |
| Presenteeism | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | ·C/O | | | |
| | Valid N | 0 | | | |
| | N missing | | | | |
| Work productivity loss | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Activity Impairment / disability | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |

Table 24. Indirect health care – Ad-hoc questionnaire (secondary objective 6)

| | | NT1 | NT2 | Total | p-value |
|---|---|---|---|---|---|
| Days off work (sick leave) in the last year | Mean (SD) | | | | |
| due to narcolepsy, n (%) | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |

Document: SAP SOMNUS

Author:


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



| | | NT1 | NT2 | Total | p-value |
|---|---|---|---|---|---|
| | Valid N (1) | | | | |
| | N missing | | | | |
| Narcolepsy has influenced/affected the fact | No | | | | |
| that you do not work, n (%) | Yes | | | | |
| | Valid N (2) | | | | |
| | N missing | | | | |
| Due to narcolepsy your level of work | No | | | | |
| productivity is or has been lower, n (%) | Yes | | | | |
| | Valid N (1) | .\ | | | |
| | N missing | 17 | | | |
| Narcolepsy has affected you or may have | No | | | | |
| affected your lack of professional promotion, n (%) | Yes | | | | |
| promotion, if (70) | Valid N (1) | | | | |
| | N missing | | | | |
| Near miss accidents, n (%) | No | | | | |
| | Yes | | | | |
| | Related with symptoms | | | | |
| | Due to medications | | | | |
| | Other | | | | |
| 1.0 <sup>X</sup> | Required ambulance presence | | | | |
| X | Required ER Visit | | | | |
| | Required Hospital Admission | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Motor vehicle accidents, n (%) | No | | | | |
| | Yes | | | | |
| | Related with symptoms | | | | |
| | Due to medications | | | | |
| | Other | | | | |
| | Required ambulance presence | | | | |
| | Required ER Visit | | | | |
| | Required Hospital Admission | | | | |

Document: SAP SOMNUS


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



| | | NT1 | NT2 | Total | p-value |
|---|---|---|---|---|---|
| | Valid N | | | | |
| | N missing | | | | |
| Work-related accident, n (%) | No | | | | |
| | Yes | | | | |
| | Related with symptoms | | | | |
| | Due to medications | | | | |
| | Other | | | | |
| | Required ambulance presence | | | | |
| | Required ER Visit | 1 | | | |
| | Required Hospital Admission | 7 | | | |
| | Valid N | | | | |
| | N missing | | | | |

<sup>(1)</sup> Patients who have worked

# Healthcare resources before diagnosis of narcolepsy 18.6.2

Utilization of health care resources associated with narcolepsy before diagnosis -Table 25. outpatients visits (exploratory objective 3)

| | | NT1 | NT2 | Total | p-value |
|---|---|---|---|---|---|
| Routine monitoring visits, n (%) | No | | | | |
| | Yes | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Total number of routine monitoring | Mean (SD) | | | | |
| visits | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Specialists involved, n (%) | Total | | | | |

Document: SAP SOMNUS


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015

<sup>(2)</sup> Patients who have not worked in the last year



| | | NT1 | NT2 | Total | p-value |
|---|---|---|---|---|---|
| | General Practitioner | | | | |
| | Specialist | | | | |
| | Neurologist | | | | |
| | Neurophysiologist | | | | |
| | Psychiatrist | | | | |
| | Other | | | | |
| | Other 1 | | | | |
| | Valid N | \ | | | |
| | N missing | 10/2 | | | |
| Number of visits to General | Mean (SD) | 0, | | | |
| Practitioner | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Number of visits to Neurologist | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid | | | | |
| | Nmissing | | | | |
| Number of visits to | Mean (SD) | | | | |
| Neurophysiologist | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Number of visits to Psychiatrist | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Number of visits to other specialist | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |

Document: SAP SOMNUS


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



| | NT1 | NT2 | Total | p-value |
|-----------|-----|-----|-------|---------|
| Min-Max | | | | |
| Valid N | | | | |
| N missing | | | | |

Table 26. Utilization of health care resources associated with narcolepsy before diagnosis – Tests conducted (exploratory objective 3)

| | | NT1 | NT2 | Total | p-value |
|---|---|---|---|---|---|
| Tests, n (%) | No | | | | |
| | Yes | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Total number of tests | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Tests conducted, n (%) | Clinical history | | | | |
| | Presence of cataplexy | | | | |
| | Neurological Assessment | | | | |
| | Clinical Assessment | | | | |
| | Determination of Hypocretin-1 CSF or Orexin | | | | |
| | Apnea-hypopnea index (AHI) | | | | |
| | Number of sleep-onset REM periods (SOREMPs) | | | | |
| | ESS | | | | |
| | PSG | | | | |
| | MSLT | | | | |
| | Laboratory | | | | |
| | Other | | | | |
| | Other 1 | | | | |
| | | | | - | |
| | Valid N | | | | |

Document: SAP SOMNUS


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



| | | NT1 | NT2 | Total | p-value |
|---|---|---|---|---|---|
| | N missing | | | | |
| Number of clinical histories | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Number of Presence of cataplexy | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Number of Neurological Assessment | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Number of Clinical Assessment | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Number of Determination of | Mean (SD) | | | | |
| Hypocretin-1 CSF or Orexin | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Number of Apnea-hypopnea index | Mean (SD) | | | | |
| (AHI) | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| | Mean (SD) | | | | |
| | ` ' | | 1 | | 1 |

Document: SAP SOMNUS


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



| | | NT1 | NT2 | Total | p-value |
|---|---|---|---|---|---|
| Number of Number of sleep-onset | Median (Q1-Q3) | | | | |
| REM periods (SOREMPs) | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Number of ESS | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Number of PSG | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Number of MSLT | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Number of laboratories | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Number of Other | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |

Table 27. Utilization of health care resources associated with narcolepsy before diagnosis –

| Emergenc | y visits (exploratory objective 3) |
|---|---|
| Document: | SAP SOMNUS |

Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



| | | NT1 | NT2 | Total | p-value |
|---|---|---|---|---|---|
| Emergency visits, n (%) | No | | | | |
| | Yes | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Total number of emergency visits | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | 1 | | |

Table 28. Utilization of health care resources associated with narcolepsy before diagnosis – Hospitalizations (exploratory objective 3)

| | | NTI | NT2 | Total | p-value |
|---|---|---|---|---|---|
| Hospitalizations, n (%) | No | No | | | |
| | Yes | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Total number of Hospitalizations | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Hospitalizations durations (days) | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |

Table 29. Utilization of health care resources associated with narcolepsy before diagnosis – complications derived from narcolepsy (exploratory objective 3)

Document: SAP SOMNUS


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



| | | NT1 | NT2 | Total | p-value |
|---|---|---|---|---|---|
| Complications, n (%) | No | | | | |
| | Yes | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Total number of complications | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | 1 | | | |
| Type of complications, n (%) | Obesity | <i>U</i> , | | | |
| | Interference with intimate relationships | | | | |
| | Fertility | | | | |
| | Physical harm: Attending to psychiatrist | | | | |
| | Work problems | | | | |
| | Others | | | | |
| | Other 1 | | | | |
| | Valid N | | | | |
| | N missing | | | | |

# 18.7 Patient Reported Outcomes (PRO)

#### 18.7.1 Health-Related Quality of Life (HRQoL)

Table 30. EQ-5D Questionnaire (secondary objective 7)

| | | NT1 | NT2 | Total | p-value |
|---|---|---|---|---|---|
| Mobility, n (%) | I have no problems in walking about | | | | |
| | I have slight problems in walking about | | | | |
| | I have moderate problems in walking about | | | | |
| | I have severe problems in walking about | | | | |
| | I am unable to walk about | | | | |
| | Valid N | | | | |

Document: SAP SOMNUS


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



| | | NT1 | NT2 | Total | p-value |
|---|---|---|---|---|---|
| | N missing | | | | |
| Self-Care, n (%) | I have no problems washing or dressing myself | | | | |
| | I have slight problems washing or dressing myself | | | | |
| | I have moderate problems washing or dressing myself | | | | |
| | I have severe problems washing or dressing myself | | | | |
| | I am unable to wash or dress myself | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Usual activities, n (%) | I have no problems doing my usual activities | | | | |
| | I have slight problems doing my usual activities | | | | |
| | I have moderate problems doing my usual activities | | | | |
| | I have severe problems doing my usual activities | | | | |
| | I am unable to do my usual activities | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Pain / Discomfort, n (%) | I have no pain or discomfort | | | | |
| | I have slight pain or discomfort | | | | |
| | I have moderate pain or discomfort | | | | |
| | I have severe pain or discomfort | | | | |
| | I have extreme pain or discomfort | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Anxiety / Depression, n | I am not anxious or depressed | | | | |
| (%) | I am slightly anxious or depressed | | | | |
| | I am moderately anxious or depressed | | | | |
| | I am severely anxious or depressed | | | | |
| | I am extremely anxious or depressed | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| EQ VAS (0-100) | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |

Document: SAP SOMNUS


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



| | NT1 | NT2 | Total | p-value |
|-----------|-----|-----|-------|---------|
| Valid N | | | | |
| N missing | | | | |

#### 18.7.2 Perception of stigma

Table 31. Description of SSCI score (secondary objective 8)

| | | NT1 | NT2 | Total | p-value |
|----------------------|----------------|------|-----|-------|---------|
| SSCI-8 score | Mean (SD) | | | \ | |
| | Median (Q1-Q3) | | | 9/3 | |
| | Min-Max | | | )` | |
| | Valid N | | S | | |
| | N missing | | . 2 | | |
| SSCI-8 | = 8 points | 4 | Clo | | |
| (categorical), n (%) | > 8 points | 20 | | | |
| | Valid N | JII. | | | |
| | N missing | 60/ | | | |

#### Treatment satisfaction 18.7.3

Description of TSQM-9 domains score (secondary objective 9) Table 32.

| | | NT1 | NT2 | Total | p-value |
|---------------|----------------|-----|-----|-------|---------|
| Effectiveness | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Convenience | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |

Document: SAP SOMNUS

Author: Version Number: 1.0 Version Date:

[19JAN2023]

Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



| | | NT1 | NT2 | Total | p-value |
|---------------------|----------------|-----|-----|-------|---------|
| | N missing | | | | |
| Global satisfaction | Mean (SD) | | | | |
| | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |

# 18.8 Factors related to healthcare resources utilization, quality of life, stigma and satisfaction

Table 33. Multivariate linear regression analysis of the sociodemographic and clinical characteristics related to healthcare resources utilization - number of routine monitoring visits in the last year

| Variable | | Univariate | Multivariate* | | | |
|---|---|---|---|---|---|---|
| | | Pr> t | Estimate | Standard<br>error | t-value | Pr> t |
| Intercept | <c< td=""><td>-</td><td></td><td></td><td></td><td></td></c<> | - | | | | |
| Age | | | | | | |
| Gender | | | | | | |

<sup>\*</sup> variables with p<0.1 in the univariate

Table 34. Multivariate linear regression analysis of the sociodemographic and clinical characteristics related to healthcare resources utilization - number of tests conducted in the last year

Document: SAP SOMNUS
Author:


Reference: RWI\_WI\_BIOS0015

Effective Date: 15Oct2021

Template No.: RWI\_TP\_BIOS0013 Revision 2



| Variable | Univariate | | Multivariate* | | |
|-----------|------------|----------|-------------------|---------|-------|
| | Pr> t | Estimate | Standard<br>error | t-value | Pr> t |
| Intercept | - | | | | |
| Age | | | | | |
| Gender | | | | | |

<sup>\*</sup> variables with p<0.1 in the univariate

Table 35. Multivariate linear regression analysis of the sociodemographic and clinical characteristics related to healthcare resources utilization - number of emergency visits in the last year

| Vari | able | Univariate | Multivariate* | | | |
|---|---|---|---|---|---|---|
| | | Przfi | Estimate | Standard<br>error | t-value | Pr> t |
| Intercept | | - 17 - | | | | |
| Age | < | | | | | |
| Gender | | | | | | |

<sup>\*</sup> variables with p<0.1 in the univariate

Table 36. Multivariate linear regression analysis of the sociodemographic and clinical characteristics related to healthcare resources utilization - number of hospitalizations in the last year

Document: SAP SOMNUS

Author: Version Number:


1.0

Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



| Variable | Univariate | | Multivariate* | | |
|-----------|------------|----------|-------------------|---------|-------|
| | Pr> t | Estimate | Standard<br>error | t-value | Pr> t |
| Intercept | - | | | | |
| Age | | | | | |
| Gender | | | | | |

Table 37. Multivariate linear regression analysis of the sociodemographic and clinical characteristics related to healthcare resources utilization number of complications in the last year

| Variable | Univariate | Multivariate* | | | |
|---|---|---|---|---|---|
| | Pr> t | Estimate | Standard<br>error | t-value | Pr> t |
| Intercept | 001 - | | | | |
| Age | o's | | | | |
| Gender | | | | | |

Table 38. Multivariate linear regression analysis of the sociodemographic and clinical characteristics related to QoL – EQ VAS

| Variable | Univariate | Multivariate* | |
|-----------|------------|---------------|------------------------|
| | Pr> t | Estimate | Standard t-value Pr> t |
| Intercept | - | | |

Document: SAP SOMNUS

Author:


1.0


. . .

Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



| Variable | Univariate | Multivariate* | | | |
|----------|------------|---------------|-------------------|---------|-------|
| | Pr> t | Estimate | Standard<br>error | t-value | Pr> t |
| Age | | | | | |
| Gender | | | | | |

Table 39. Multivariate linear regression analysis of the sociodemographic and clinical characteristics related to stigma – SSCI-8 score

| Variable | Univariate | 1150 | Multivariate* | | |
|-----------|----------------|-------------|---------------|---------|-------|
| | Pr> t | Estimate | Standard | t-value | Pr> t |
| | e C | () <b>`</b> | error | | |
| Intercept | - 011 | | | | |
| Age | CO, | | | | |
| Gender | 2011 | | | | |
| | o <sup>r</sup> | | | | |

Table 40. Multivariate linear regression analysis of the sociodemographic and clinical characteristics related to stigma – TSQM-9 global satisfaction score

| Variable | Univariate | Multivariate* | | | |
|-----------|------------|---------------|-------------------|---------|-------|
| | Pr> t | Estimate | Standard<br>error | t-value | Pr> t |
| Intercept | - | | | | |
| Age | | | | | |
| Gender | | | | | |

Document: SAP SOMNUS

Author:


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



| Variable | Univariate | Multivariate* | | | |
|----------|------------|---------------|-------------------|---------|-------|
| | Pr> t | Estimate | Standard<br>error | t-value | Pr> t |

# 18.9 Proportion of patients with narcolepsy diagnosed and managed in public hospitals

Table 41. Patients with narcolepsy (with and without cataplexy) diagnosed and managed in public hospitals (exploratory objective 1)

| Only public hospitals | | Total | Type 1 | Type 2 |
|---|---|---|---|---|
| Total population under the hospital's | Mean (SD) | | - | - |
| circumscription | Median (Q1-Q3) | | - | - |
| | Min-Max | | - | - |
| | Valid N | | - | - |
| | N missing | | - | - |
| Total of patients with narcolepsy | Mean (SD) | | | |
| attended in the participating site according to routine clinical practice | Median (Q1-Q3) | | | |
| and type of narcolepsy | Min-Max | | | |
| | Valid N | | | |
| | N missing | | | |
| Proportion of patients with narcolepsy | (%) | | | |
| New patients with narcolepsy diagnosed | Mean (SD) | | | |
| per year | Median (Q1-Q3) | | | |
| | Min-Max | | | |
| | Valid N | | | |
| | N missing | | | |
| Proportion of new patients with narcolepsy | (%) | | | |

Document: SAP SOMNUS

Author:


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



# 18.10 Sociodemographic and clinical characteristics of patients with narcolepsy according to treated and untreated patients.

Following tables will be analyzed considering the type of narcolepsy (NT1 and NT2)

Table 42. Sociodemographic and clinical characteristics of patients with narcolepsy stratified by treated and untreated patients (secondary objective 1)

| | | Untreated (naïve) | Treated | Total | p-value |
|---|---|---|---|---|---|
| Age at the time of the visit, | Mean (SD) | , | | | |
| years | Median (Q1-Q3) | | | | |
| | Min-Max | | 3 | | |
| | Valid N | 0, | | | |
| | N missing | 50 | | | |
| Gender, n (%) | Male | V. | | | |
| | Female | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Ethnicity, n (%) | Caucasian | | | | |
| | Hispanic | | | | |
| | African | | | | |
| | Asian / Oriental | | | | |
| | Other | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Educational level ongoing or | Without studies | | | | |
| completed level of education, n (%) | Primary Studies | | | | |
| (70) | Secondary Studies | | | | |
| | University Studies | | | | |
| | Other Superior Studies | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Occupational status and | Student | | | | |
| occupation, n (%) | Employed | | | | |

Document: SAP SOMNUS


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



| | | Untreated (naïve) | Treated | Total | p-value |
|---|---|---|---|---|---|
| | Self-employed | | | | |
| | Employed but on sick leave due to the study disease | | | | |
| | Permanent incapacity to work due to the study disease | | | | |
| | Permanent incapacity to work due to other reasons | | | | |
| | Unemployed | | | | |
| | Retired | | | | |
| | Domestic work | | 1 | | |
| | Other | 20 | | | |
| | Valid N | 0, | | | |
| | N missing | 115 | | | |
| Civil status, n (%) | Married/with partner | <u> </u> | | | |
| | Divorced/separated | | | | |
| | Unmarried | | | | |
| | Widow/er | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Living conditions, n (%) | Alone | | | | |
| | Wife/Husband and /or sons | | | | |
| | Family Caregivers | | | | |
| | Other Caregivers | | | | |
| | Valid N | | | | |
| | N missing | | | | |

Table 43. Patients' physical examination at study visit stratified by treated and untreated patients (secondary objective 1)

| | | Untreated (naïve) | Treated | Total | p-value |
|----|----------------|-------------------|---------|-------|---------|
| Me | Iean (SD) | , | | | |
| Me | Iedian (Q1-Q3) | | | | |

Document: SAP SOMNUS

Author:


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



| | | Untreated (naïve) | Treated | Total | p-value |
|---|---|---|---|---|---|
| Height at treatment start or last | Min-Max | | | | |
| available before treatment | Valid N | | | | |
| initiation, cm | N missing | | | | |
| Weight at treatment start or last | Mean (SD) | | | | |
| available before treatment initiation, kg | Median (Q1-Q3) | | | | |
| minution, kg | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| BMI, kg/m <sup>2</sup> | Mean (SD) | 2 | 3 | | |
| | Median (Q1-Q3) | 0/ | | | |
| | Min-Max | 50 | | | |
| | Valid N | 0 | | | |
| | N missing | | | | |
| Blood pressure (systolic), | Mean (SD) | | | | |
| mmHg | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Blood pressure (diastolic), | Mean (SD) | | | | |
| mmHg | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Smoking status, n(%) | Current Smoker | | | | |
| | Ex-Smoker | | | | |
| | Non-Smoker | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Alcohol intake, n(%) | Never | | | | |
| | Once or less per month | | | | |
| | 2-4 times per month | | | | |

Document: SAP SOMNUS


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



| | | Untreated (naïve) | Treated | Total | p-value |
|---|---|---|---|---|---|
| | 2-3 times per week | | | | |
| | 4 or more times per week | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Exercise status, n(%) | Never | | | | |
| | Regular (1 - 3times/week) | | | | |
| | Frequently (4 - 7 times /week) | | | | |
| | Always (7 or more times/week) | | 4 | | |
| | Valid N | 2 | 7 | | |
| | N missing | 0/ | | | |
| Family history of narcolepsy in | No | 50 | | | |
| first- or second-degree relatives, n (%) | Yes | | | | |
| 101dt1 v 03, 11 (70) | First-degree relatives | | | | |
| | Second-degree relatives | | | | |
| | Valid N | | | | |
| | N missing | | | | |

# 18.11 Adverse drug reaction associated to narcolepsy treatments

Table 44. Adverse events (AE) associated to narcolepsy treatments (secondary objective 11)

| | | Adverse even | Adverse event related to a Takeda produc | |
|---|---|---|---|---|
| | | No | Yes | Total |
| Adverse event, n (%) | No | | | |
| | Yes | | | |
| | Valid N | | | |
| | N missing | | | |
| Type of AE* | SOC1 | | | |
| | PT1 | | | |

Document: SAP SOMNUS


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



| | Adverse event related to a Takeda produc | | |
|-----------|------------------------------------------|-----|-------|
| | No | Yes | Total |
| SOC2 | | | |
| PT1 | | | |
| Valid N | | | |
| N missing | | | |

<sup>\*</sup>MedDRA codification

#### 19. ANNEX

All those tables presented in section 18 of this document and that are stratified by type of narcolepsy will be analyzed in addition to type of narcolepsy by type of center (public or private). These tables will be included in an annex to the statistical.

The following two tables are shown as an example:

Table 45. Patients' sociodemographic and baseline characteristics by type of center (NT1)

| | | NT1 | | Total | p- |
|---|---|---|---|---|---|
| | | Public | Private | | value |
| Age at the time of the visit, | Mean (SD) | | | | |
| years | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Gender, n (%) | Male | | | | |
| | Female | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Ethnicity, n (%) | Caucasian | | | | |

Document:

SAP SOMNUS

Template No.: RWI\_TP\_BIOS0013 Revision 2

Author:


1.0


Reference: RWI\_WI\_BIOS0015



| | | NT1 | | Total | |
|---|---|---|---|---|---|
| | | Public | Private | 1 | value |
| | Hispanic | | | | |
| | African | | | | |
| | Asian / Oriental | | | | |
| | Other | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Educational level ongoing or | Without studies | | | | |
| completed level of education, n (%) | Primary Studies | | | | |
| (70) | Secondary Studies | | | | |
| | University Studies | | | | |
| | Other Superior Studies | | | | |
| | No available | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Occupational status and | Student | | | | |
| occupation, n (%) | Employed | | | | |
| | Self-employed | | | | |
| | Employed but on sick leave due to the study disease | | | | |
| | Permanent incapacity to work due to the study disease | | | | |
| | Permanent incapacity to work due to other reasons | | | | |
| | Unemployed | | | | |
| | Retired | | | | |
| | Domestic work | | | | |
| | Other | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Civil status, n (%) | Married/with partner | | | | |
| | Divorced/separated | | | | |
| | Unmarried | | | | |
| | Widow/er | | | | |

Document: SAP SOMNUS


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



| | | NT1 | | Total | p- |
|---|---|---|---|---|---|
| | | Public | Private | | value |
| | Valid N | | | | |
| | N missing | | | | |
| Living conditions, n (%) | Alone | | | | |
| | Wife/Husband and /or sons | | | | |
| | Family Caregivers | | | | |
| | Other Caregivers | | | | |
| | Valid N | | | | |
| | N missing | | | | |

Table 46. Patients' sociodemographic and baseline characteristics by type of center (NT2)

| | | N | T2 | Total | ıl p-<br>value |
|---|---|---|---|---|---|
| | Mercie | Public | Private | 1 | |
| Age at the time of the visit, | Mean (SD) | | | | |
| years | Median (Q1-Q3) | | | | |
| | Min-Max | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Gender, n (%) | Male | | | | |
| | Female | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Ethnicity, n (%) | Caucasian | | | | |
| | Hispanic | | | | |
| | African | | | | |
| | Asian / Oriental | | | | |
| | Other | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| | Without studies | | | | |

Document: SAP SOMNUS


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



| | | NT2 | | Total | |
|---|---|---|---|---|---|
| | | Public | Private | | value |
| Educational level ongoing or completed level of education, n | Primary Studies | | | | |
| | Secondary Studies | | | | |
| | University Studies | | | | |
| | Other Superior Studies | | | | |
| (%) | No available | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Occupational status and | Student | | | | |
| occupation, n (%) | Employed | | | | |
| | Self-employed | | | | |
| | Employed but on sick leave due to the study disease | | | | |
| | Permanent incapacity to work due to the study disease | | | | |
| | Permanent incapacity to work due to other reasons | | | | |
| | Unemployed | | | | |
| | Retired | | | | |
| | Domestic work | | | | |
| | Other | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Civil status, n (%) | Married/with partner | | | | |
| | Divorced/separated | | | | |
| | Unmarried | | | | |
| | Widow/er | | | | |
| | Valid N | | | | |
| | N missing | | | | |
| Living conditions, n (%) | Alone | | | | |
| | Wife/Husband and /or sons | | | | |
| | Family Caregivers | | | | |
| | Other Caregivers | | | | |
| | Valid N | | | | |

Document: SAP SOMNUS


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015



| | N | NT2 | p- |
|-----------|--------|---------|-------|
| | Public | Private | value |
| N missing | | | |

For non-commercial use only

Document: SAP SOMNUS


Template No.: RWI\_TP\_BIOS0013 Revision 2 Reference: RWI\_WI\_BIOS0015